CLINICAL TRIAL: NCT01945996
Title: Trial to Examine Text-based mHealth for Emergency Department Patients With Diabetes With Family And Friend Network Supporter
Brief Title: Harnessing mHealth and Social Support to Improve Diabetes Related Health Behavior for Inner-city Patients
Acronym: TExTMEDFANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Elizabeth Burner, Assistant Professor of Clinical Emergency Medicine, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HS-13-00382; KL2TR000131 (NIH)
Record Dates: First submitted 2013-08-30; First posted 2013-09-19 (Estimated); Results first posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus
Keywords: Hispanic Americans; Cellular Phone; Behavior
MeSH Terms: conditions — Diabetes Mellitus; Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- TExT-MED only (Active Comparator): Patients will receive TExT-MED intervention, but supporters will not receive additional messages
  Interventions: Behavioral: TExT MED
- TExT-MED FANS (Experimental): Patients get TExT-MED intervention, supporter gets FANS curriculum
  Interventions: Behavioral: TExT MED; Behavioral: FANS

INTERVENTIONS:
Behavioral: TExT MED — educational , motivational, medication reminder and healthy living challenge text messages sent to patient's cell phone
Behavioral: FANS — supporter curriculum of messages, consisting of educational/motivational messages, and support challenges
  Arms: TExT-MED FANS

SUMMARY:
In this study, an existing mobile health intervention to improve diabetes self-management will be combined with a social support module and tested for feasibility. The investigators hypothesize that this combination will be feasible and acceptable to both patients and their loved ones.

DETAILED DESCRIPTION:
This will be the first ever evaluation of a highly scalable and low-cost social support intervention for patients with diabetes delivered entirely via mobile phones. TExT-MED FANS (Trial to Examine Text-based mHealth for Emergency Department Patients With Diabetes With Family And Friend Network Supporter) will unite the benefits of mHealth (scalability, ease of access) and social support interventions (personalized motivation, emotional support). The Diabetes FANS text message based curriculum will make it easier for friends and family to become supporters. Additionally, augmenting TExT-MED with the FANS social support module will be more effective than TExT-MED alone. The personalized support of TExT-MED FANS will also be more effective than providing TExT-MED in combination with a community health worker supporter who lacks a pre-existing relationship with the patient. Through this innovative combination, I can create a more cost-effective and diffusible mHealth solution that maintains the personal connection of social support interventions. To date there has only been one study evaluating social support interventions for patients with diabetes using mHealth, but in this study participants were paired with other subjects with diabetes (not friends or family) and it required intensive face-to-face support group time. TExT-MED FANS will provide key insights into the utility of combining social support interventions delivered solely via mHealth in low-income Latino patients. These insights will help future interventions achieve maximal impact on diabetes and other chronic disease management.

ELIGIBILITY:
Inclusion Criteria:

* type II diabetes
* HbA1c >or=8 at enrollment
* speak English or Spanish
* has support person willing to participate

Exclusion Criteria:

* unable to consent
* pediatric patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- LAC+USC, Los Angeles, California, United States

REFERENCES:
- [Background] Burner E, Menchine M, Taylor E, Arora S. Gender differences in diabetes self-management: a mixed-methods analysis of a mobile health intervention for inner-city Latino patients. J Diabetes Sci Technol. 2013 Jan 1;7(1):111-8. doi: 10.1177/193229681300700113. PMID 23439166
- [Background] Arora S, Peters AL, Agy C, Menchine M. A mobile health intervention for inner city patients with poorly controlled diabetes: proof-of-concept of the TExT-MED program. Diabetes Technol Ther. 2012 Jun;14(6):492-6. doi: 10.1089/dia.2011.0252. Epub 2012 Apr 23. PMID 22524591

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 745 patients screened
  Excluded:
  * No mobile phone = 174
  * Do not know how to text = 180
  * HbA1c <8 = 145
  * No English or Spanish = 28
  * Critically ill/AMS = 80
  * Refused screening = 28
Pre-assignment Details: 14 patients dropped before randomization
  * Unable to identify support person = 4
  * Unable to contact support person = 22
  * Support person can not text = 15
Groups:
- TExT-MED Only: Patients will receive TExT-MED (Trial to Examine Text-Based mHealth for Emergency department patients with Diabetes) intervention, but supporters will not receive additional messages
  TExT MED: educational , motivational, medication reminder and healthy living challenge text messages sent to patient's cell phone
- TExT-MED FANS: Patients get TExT-MED intervention, supporter gets FANS curriculum (Trial to Examine Text-Based mHealth for Emergency department patients with Diabetes with Family And friends Network Supporters)
  TExT MED: educational , motivational, medication reminder and healthy living challenge text messages sent to patient's cell phone
  FANS: supporter curriculum of messages, consisting of educational/motivational messages, and support challenges
Period: Overall Study
Arm/Group | TExT-MED Only | TExT-MED FANS
Started | 22 | 22
Completed | 19 | 17
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TExT-MED Only | TExT-MED FANS | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.05 (9.17) | 46.04 (9.86) | 46.05 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 8 | 11 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-hispanic White | 1 | 1 | 2
  Latino | 18 | 17 | 35
  African American | 2 | 1 | 3
  Asian | 1 | 1 | 2
  Other | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 22 | 44
Language [Count of Participants; unit: Participants]
  Both Equally | 1 | 1 | 2
  More English than Spanish | 2 | 4 | 6
  More Spanish than English | 4 | 3 | 7
  Only English | 2 | 2 | 4
  Only Spanish | 11 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Feasibility
Description: Number of patients lost to follow-up
Time Frame: 3 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | TExT-MED Only | TExT-MED FANS
Number analyzed (Participants) | 22 | 22
Participants | 3 | 5

2. Primary Outcome: Acceptability
Description: Patient response to: I have enjoyed the TExT-MED FANS (Trial to Examine Text-based mHealth for Emergency Department Patients With Diabetes With Family And Friend Network Supporter) program?
Time Frame: 3 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | TExT-MED Only | TExT-MED FANS
Number analyzed (Participants) | 19 | 17
Participants
  Yes | 18 | 17
  No | 1 | 0

3. Primary Outcome: Acceptability 2: Would Patients Recommend the Program to Family or Friends?
Description: Response to: Would you recommend TExT-MED FANS to family or friends?
Time Frame: 3 months follow up
Measure: Count of Participants; unit: Participants
Arm/Group | TExT-MED Only | TExT-MED FANS
Number analyzed (Participants) | 19 | 17
Participants
  Yes | 18 | 17
  No | 1 | 0

4. Secondary Outcome: Diabetes Knowledge Test Scale
Description: Diabetes Knowledge Test Scale measures specific areas of diabetes knowledge, and is geared to specific curriculum
Time Frame: 3 months after enrollment
Population: Data was not collected as final program educational curriculum did not have sufficient overlap with Diabetes Knowledge Test Scale
Arm/Group | TExT-MED Only | TExT-MED FANS
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Self-efficacy
Description: Change Diabetes Empowerment Scale - Short Form( measures feelings of self efficacy regarding diabetes disease management) from baseline to 6 month follow up scale minimum 8, maximum 40 Best possible change 40 (maximum at follow up) minus 8 (minimum at follow up)=32 Worst possible change: -32
Time Frame: 3 months after enrollment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED FANS
Number analyzed (Participants) | 19 | 17
units on a scale | .3 [-.1 to 0.7] | 0.1 [-.2 to 0.4]

6. Secondary Outcome: Change in Problem Areas in Diabetes Scale
Description: Change in Problem areas in diabetes scale (a measure of mental health problems that patient experience related to their diabetes) Baseline minus 3 month follow up.
  Higher score = more problems scale minimum 0 scale maximum 100 worst possible change -100 (0 problem scale at baseline, 100 at follow up) best possible change 100 (100 problem scale at baseline, 0 at follow up
Time Frame: 3 months after enrollment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED FANS
Number analyzed (Participants) | 19 | 17
units on a scale | -.9 [-15 to 13.2] | -6.8 [-16 to -3.8]

7. Secondary Outcome: Glycemic Control
Description: glycosylated hemoglobin A1c
Time Frame: 3 months after enrollment
Measure: Mean (95% Confidence Interval); unit: % glycoslated hemoglobin
Arm/Group | TExT-MED Only | TExT-MED FANS
Number analyzed (Participants) | 19 | 17
% glycoslated hemoglobin | -0.6 [-1.4 to 0.2] | -1.4 [-2.3 to -0.4]

8. Secondary Outcome: Body Mass Index
Description: height and weight measurements
Time Frame: 3 months after enrollment
Population: Was not able to be collected
Arm/Group | TExT-MED Only | TExT-MED FANS
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Summary of Diabetes Self-care Activities - General Diet Sub Score
Description: change in number of days patient followed a general diet plan (3 month follow up report minus baseline report) Minimum -7: worst possible change (from all days at baseline to no days at follow up) Max 7: best possible change from baseline (from no days at baseline to all days at follow up)
Time Frame: 3 months follow up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED FANS
Number analyzed (Participants) | 19 | 17
units on a scale | 0.1 [-1 to 1.3] | 0.9 [-.3 to 2]

10. Secondary Outcome: Change in Summary of Diabetes Self-care Activities - Specific Diet Sub Score
Description: change in number of days patient followed a diabetes specific diet plan (3 month follow up report minus baseline report) Minimum -7: worst possible change (from all days at baseline to no days at follow up) Max 7: best possible change from baseline (from no days at baseline to all days at follow up)
Time Frame: 3 months follow up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED FANS
Number analyzed (Participants) | 19 | 17
units on a scale | 0.9 [-.1 to 1.9] | 1.2 [0.2 to 2]

11. Secondary Outcome: Change in Summary of Diabetes Self-care Activities - Exercise Sub Score
Description: change in number of days patient exercised (3 month follow up report minus baseline report) Minimum -7: worst possible change (from all days at baseline to no days at follow up) Max 7: best possible change from baseline (from no days at baseline to all days at follow up)
Time Frame: 3 months follow up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED FANS
Number analyzed (Participants) | 19 | 17
units on a scale | 0.7 [-.6 to 2] | 0.4 [-.6 to 1.3]

12. Secondary Outcome: Change in Summary of Diabetes Self-care Activities - Blood Glucose Sub Score
Description: change in number of days patient checked blood sugar (3 month follow up report minus baseline report) Minimum -7: worst possible change (from all days at baseline to no days at follow up) Max 7: best possible change from baseline (from no days at baseline to all days at follow up)
Time Frame: 3 months follow up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED FANS
Number analyzed (Participants) | 19 | 17
units on a scale | -.7 [-2 to 0.7] | 1.6 [0.5 to 2.7]

13. Secondary Outcome: Change in Summary of Diabetes Self-care Activities - Foot Care Sub Score
Description: change in number of days patient followed a foot care plan (3 month follow up report minus baseline report) Minimum -7: worst possible change (from all days at baseline to no days at follow up) Max 7: best possible change from baseline (from no days at baseline to all days at follow up)
Time Frame: 3 months follow up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED FANS
Number analyzed (Participants) | 19 | 17
units on a scale | 0.9 [-.3 to 2.1] | 1 [-.5 to 2.6]

14. Secondary Outcome: Change in Summary of Diabetes Self-care Activities - Carb Spacing Sub Score
Description: change in number of days patient followed a carb spacing plan (3 month follow up report minus baseline report) Minimum -7: worst possible change (from all days at baseline to no days at follow up) Max 7: best possible change from baseline (from no days at baseline to all days at follow up)
Time Frame: 3 months follow up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TExT-MED Only | TExT-MED FANS
Number analyzed (Participants) | 19 | 17
units on a scale | 0.5 [-.6 to 1.5] | 0.5 [-.7 to 1.6]

ADVERSE EVENTS:
Time Frame: 3 months
Description: patients reported any adverse events
Arm/Group | TExT-MED Only | TExT-MED FANS
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

LIMITATIONS AND CAVEATS:
BMI was not able to be collected. Diabetes knowledge test was removed from follow up as intervention did not teach sufficient content to overlap with scale Unable to measure actual text receipt on the mobile platform used

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No